CLINICAL TRIAL: NCT04333524
Title: FDG PET Evaluation for Marginal Zone Lymphoma and Its Prognostic Role: an International Multicenter Retrospective Analysis
Brief Title: FDG PET Evaluation for Marginal Zone Lymphoma and Its Prognostic Role
Acronym: PIMENTO
Status: Active, not recruiting | Type: Observational
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Responsible Party: Sponsor
Other Study IDs: IELSG44
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Marginal Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Staging
- Group B: Criteria for response assessment

SUMMARY:
The general aim of the present study is to assess the role of PET for the staging and for the assessment of response and outcome prediction in Marginal Zone Lymphoma (MZL). This study will be conducted as a multicenter retrospective analysis of MZL for whom PET scan are available as DICOM file for central review.

The study is designed as a retrospective collection of patients with MZL enrolled in the prospective IELSG36 and IELSG38 trials sponsored by IELSG and in the observational NF10 study sponsored by Federazione Italiana Linfomi (FIL), with the possibility to add additional cases from participating institutions.

The study will be conducted on performed scans. No additional scan or procedure will be required for study purposes.

The study will be divided into two sections with different aims:

Part A will be conducted to understand the role of PET for the staging of MZL. PET scans will be analyzed and compared with data retrieved from CT scan and from other staging procedures, also including bone marrow biopsy, ultrasound, and laboratory exams. This part of the study will describe ability of PET to identify pathologic lesions and to contribute to staging definition or to stage migration.

Part B will be conducted to validate standardized criteria for response assessment in MZL including FDG-PET among procedures and to define the prognostic role of metabolic response in MZL. For this purpose the primary endpoint for this part of the study is defined as the progression free survival. Secondary endpoint will be Overall survival, and response rate defined with conventional procedures and rate of histological transformation.

DETAILED DESCRIPTION:
A significant proportion of patients considered for this study will be retrieved from previous observational prospective clinical studies. Data on clinical presentation, treatment and follow-up will be obtained from the existing dataset of the previous protocols. For the additional cases identified from clinical practice data will be collected from patient chart. A unique study CRF will be prepared to collect all the required details.

Patients with histologically confirmed marginal zone lymphomas according to the current WHO classification are registered in the study. Moreover, patients characteristics (PS, systemic symptoms), Ann Arbor stage, laboratory parameters, serology for hepatitis C, B and human immunodeficiency virus, bone marrow aspirate and biopsy data, data on treatment start and end, chemotherapy details, final response defined according to Cheson 2014 and Matutes criteria, date of last follow-up ,occurrence of any event (relapse, progression, death) with date will be collected.

PET response will be initially coded according to local interpretation of scan report. All FDG-PET, will be then centralized to perform a blinded independent review of staging and response. Images will be centralized and examined by a panel of 3 nuclear medicine physicians that will independently review the scans. Each case will be evaluated by two reviewers. In case of discordant results a third reviewer will adjudicate the case.

Each patient enrolled in the study will be anonymized by assigning a unique identification numerical code upon registration in the study. The unique identification code will be used to record health-related data.

Anonymized PET data will be uploaded into the DICOM system by the responsible person of the site.

Anonymized health-related data will be collected in the e-CRF. At each site, the responsible of the research or a delegated person will complete the e-CRF.

Only the Study Chair and the Sponsor will have access rights for the health-related data and will be responsible for protection of the data.

ELIGIBILITY:
Inclusion Criteria:

1. One of the following subtypes of Histology confirmed Indolent non-follicular B-cell lymphoma:

   * Splenic MZL (bone marrow histology and/or splenic tissue);
   * Extranodal MZL or MALT (tissue biopsy);
   * Nodal MZL (lymph node biopsy).
2. Age over 18.
3. Availability of details on clinical presentation, treatment details and results, and on follow-up.
4. Execution of PET at diagnosis or/and at end of treatment or/and at relapse.
5. Execution of CT scan with iodine contrast medium at diagnosis and at assessment of response.
6. Patients with histologically confirmed marginal zone lymphomas according to the current WHO classification are registered in the study. Diagnosis based on tru-cut core-needle biopsies are permitted in the study.
7. Written informed consent.

Exclusion Criteria:

1. Patients with a diagnosis of Non Hodgkin Lymphoma other than MZL.
2. Scans images not available for whatever reason.
3. Cases diagnosed on fine needle aspiration cytology only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MZL enrolled in the prospective IELSG36 and IELSG38 trials and on the observational NF10, with the possibility to add additional cases from participating institutions
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between CT and PET | At baseline
  To correlate CT and PET results for stage definition

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From date of enrollment until the date of first documented progression, or last follow up, or date of death from any cause, whichever came first, assessed up to a maximum of 10 years
Duration of Response (DoR) | From date of first response to the date of relapse, or last follow up, or date of death from any cause, whichever came first, assessed up to a maximum of 10 years
  DoR is evaluated only for responding patients

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Luminari, MD, Study Chair — AUSL IRCCS - Reggio Emilia (Italy); Catherine Thieblemont, MD, Study Chair — Saint-Louis Hospital, Paris, France; Emanuele Zucca, MD, Study Chair — Oncology Institute of Southern Switzerland
Locations (25):
- France (3):
  - CHU de Dijon, Dijon
  - Saint Louis Hospital, Paris
  - IUCT Oncopole Toulouse, Toulouse
- Italy (20):
  - ASO SS. Antonio e Biagio e C. Arrigo, Alessandria, AL
  - Ospedale degli Infermi, Ponderano, BI
  - Ospedale Oncologico Businco, Cagliari, CA
  - "G. Rodolico", AOU Policlinico Vittorio Emanuele, Catania, CT
  - Fondazione IRCCS - Cà Granda Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale San Raffaele, Milan, MI
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI
  - AOU Policlinico "Paolo Giaccone", Palermo, PA
  - I.R.C.C.S. Istituto Oncologico Veneto, Padua, PD
  - Ospedale Civile Spirito Santo Pescara, Pescara, PE
  - IRCCS Centro di Riferimento Oncologico di Aviano, Aviano, PN
  - Fondazione IRCCS Policlinico S. Matteo di Pavia, Pavia, PV
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo, TO
  - A.O.U. Città della Salute e della Scienza di Torino, Torino, TO
  - A.O. Santa Maria di Terni, Terni, TR
  - Azienda Ospedaliera - Ospedale di Circolo e Fondazione Macchi di Varese, Varese, VA
  - Policlinico GB Rossi, Verona, VR
  - IRCCS Istituto Tumori "Giovanni Paolo II", Bari
  - AOU Federico II, Napoli
  - AUSL IRCCS Reggio Emilia, Reggio Emilia
- Switzerland (2):
  - Hôpiteux Universitaires de Genève (HUG), Geneva, Canton of Geneva
  - Istituto Oncologico della Svizzera Italiana, Bellinzona, Canton Ticino